CLINICAL TRIAL: NCT00592228
Title: Deferral of Angioplasty According to Fractional Flow Reserve vs. Routine Drug-eluting Stent Implantation in Intermediate Coronary Stenosis
Brief Title: Proper Fractional Flow Reserve Criteria for Intermediate Lesions in the Era of Drug-eluting Stent
Acronym: DEFER-DES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to slow enrollment
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Bon-Kwon Koo, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-0706-026-210
Record Dates: First submitted 2007-12-17; First posted 2008-01-11 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2010-12

CONDITIONS: Coronary Angiography; Drug-eluting Stents; Fractional Flow Reserve, Myocardial
Keywords: intermediate lesion; drug-eluting stent; fractional flow reserve

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Fractional flow guided drug-eluting stent implantation arm
  Interventions: Device: Cypher, Taxus or Endeavor
- 2 (Other): Routine drug-eluting stent implantation
  Interventions: Device: Cypher, Taxus or Endeavor

INTERVENTIONS:
Device: Cypher, Taxus or Endeavor — percutaneous drug-eluting stent implantation,
  1. FFR group: if FFR<0.75
  2. Routine DES group

SUMMARY:
Angiographic evaluation for intermediate lesions is not always accurate. Fractional flow reserve-guided deferral strategy for these lesions showed the same event rate as routine intervention strategy. However, proper FFR criterion for these lesions in the era of drug-eluting stent is not known. This study sought to evaluate the clinical outcomes of intermediate lesions according to FFR and compare those of FFR-guided intervention with routine drug-eluting stent implantation strategy.

ELIGIBILITY:
Inclusion Criteria:

* Elective PCI
* Angiographically intermediate stenosis (50-75% by visual estimation) in native major coronary arteries, proximal and mid (branch, distal lesion: exclusion)
* Reference diameter > 2.5mm, lesion length < 60mm (cover by 2 stents)
* No documented evidence of ischemia by noninvasive tests

Exclusion Criteria:

* Acute ST elevation MI
* Left main disease
* Chronic renal failure (cr >2 mg/dL)
* Expected survival < 2yrs
* > 1degree AV block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-01 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Clinical event: Cardiac death, myocardial infarction, target lesion revascularization | 9 months

SECONDARY OUTCOMES:
IVUS | at the time of procedure
  IVUS minimum lumen area

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul national university hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park SH, Jeon KH, Lee JM, Nam CW, Doh JH, Lee BK, Rha SW, Yoo KD, Jung KT, Cho YS, Lee HY, Youn TJ, Chung WY, Koo BK. Long-Term Clinical Outcomes of Fractional Flow Reserve-Guided Versus Routine Drug-Eluting Stent Implantation in Patients With Intermediate Coronary Stenosis: Five-Year Clinical Outcomes of DEFER-DES Trial. Circ Cardiovasc Interv. 2015 Dec;8(12):e002442. doi: 10.1161/CIRCINTERVENTIONS.115.002442. PMID 26643736